CLINICAL TRIAL: NCT02097966
Title: A Multicenter Compassionate Use Program of Daclatasvir (BMS-790052) in Combination With Sofosbuvir With or Without Ribavirin for the Treatment of Subjects With Chronic Hepatitis C
Brief Title: EU: A Multicenter Compassionate Use Program of Daclatasvir (BMS-790052) in Combination With Sofosbuvir With or Without Ribavirin for the Treatment of Subjects With Chronic Hepatitis C
Status: No longer available | Type: Expanded Access
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: AI444-237
Record Dates: First submitted 2014-03-25; First posted 2014-03-27 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2015-11

CONDITIONS: Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — daclatasvir; Sofosbuvir; Ribavirin

INTERVENTIONS:
Drug: Daclatasvir
  Other Names: BMS-790052
Drug: Sofosbuvir
Drug: Ribavirin

SUMMARY:
The primary objective of this program is to provide Daclatasvir in combination with Sofosbuvir with or without Ribavirin to subjects with chronic Hepatitis C who are at a high risk of liver decompensation or death within 12 months if left untreated and who have no available therapeutic options.

ELIGIBILITY:
This program is conducted in the EU (Germany, Austria, Norway, The Netherlands, Sweden and United Kingdom only)

For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Patients chronically infected with Hepatitis C
* Patients at a high risk of liver decompensation or death within 12 months if left untreated and who have no available therapeutic options

Exclusion Criteria:

* Patients who are <18 years old
* Patients who have contraindications to either Daclatasvir (DCV) or Sofosbuvir (SOF)
* Patients who are pregnant
* Creatinine clearance (CrCl) ≤ 30 mL/min (as estimated by Cockcroft and Gault formula)
* Patients who are pregnant or Women of Child Bearing Potential who are not using required contraception

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (56):
- Austria (9):
  - Local Institution, Amstetten
  - Local Institution, Braunua/Inn
  - Local Institution, Graz
  - Local Institution, Innsbruck
  - Local Institution, Linz
  - Local Institution, Oberndorf
  - Local Institution, Oberpullendorf
  - Local Institution, Salzburg
  - Local Institution, Vienna
- Germany (21):
  - Local Institution, Aachen
  - Local Institution, Augsburg
  - Local Institution, Berlin
  - Local Institution, Bonn
  - Local Institution, Cologne
  - Local Institution, Essen
  - Local Institution, Frankfurt
  - Local Institution, Frankfurt am Main
  - Local Institution, Hamburg
  - Local Institution, Hanover
  - Local Institution, Heidelberg
  - Local Institution, Herne
  - Local Institution, Jena
  - Local Institution, Kiel
  - Local Institution, Leipzig
  - Local Institution, München
  - Local Institution, Münster
  - Local Institution, Stuttgart
  - Local Institution, Tübingen
  - Local Institution, Ulm
  - Local Institution, Würzburg
- Netherlands (3):
  - Local Institution, Amsterdam
  - Local Institution, Rotterdam
  - Local Institution, Urecht
- Sweden (8):
  - Local Institution, Falun
  - Local Institution, Gothenburg
  - Local Institution, Helsingborg
  - Local Institution, Kalmar
  - Local Institution, Luleå
  - Local Institution, Lund
  - Local Institution, Stockholm
  - Local Institution, Sundsvall
- United Kingdom (15):
  - Local Institution, Plymouth, Devon
  - Local Institution, London, Greater London
  - Local Institution, Manchester, Greater Manchester
  - Local Instituition, Liverpool, Merseyside
  - Local Institution, Nottingham, Nottinghamshire
  - Local Institution, Oxford, Oxfordshire
  - Local Institution, Newcastle upon Tyne, Tyne and Wear
  - Local Institution, Birmingham, West Midlands
  - Local Institution, Leeds, Yorkshire
  - Local Institution, Brighton
  - Local Institution, Cardiff
  - Local Institution, Frimley
  - Local Institution, Guildford
  - Local Institution, London
  - Local Institution, Wrexham

REFERENCES:
- [Derived] Rockstroh JK, Ingiliz P, Petersen J, Peck-Radosavljevic M, Welzel TM, Van der Valk M, Zhao Y, Jimenez-Exposito MJ, Zeuzem S. Daclatasvir plus sofosbuvir, with or without ribavirin, in real-world patients with HIV-HCV coinfection and advanced liver disease. Antivir Ther. 2017;22(3):225-236. doi: 10.3851/IMP3108. Epub 2016 Nov 15. PMID 27845298
- [Derived] Welzel TM, Petersen J, Herzer K, Ferenci P, Gschwantler M, Wedemeyer H, Berg T, Spengler U, Weiland O, van der Valk M, Rockstroh J, Peck-Radosavljevic M, Zhao Y, Jimenez-Exposito MJ, Zeuzem S. Daclatasvir plus sofosbuvir, with or without ribavirin, achieved high sustained virological response rates in patients with HCV infection and advanced liver disease in a real-world cohort. Gut. 2016 Nov;65(11):1861-1870. doi: 10.1136/gutjnl-2016-312444. Epub 2016 Sep 7. PMID 27605539
- See also: EAP Investigator Requests — http://www.bms.com/clinical_trials/investigator_sponsored_research/Pages/expanded-access-program.aspx
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx